CLINICAL TRIAL: NCT05146544
Title: Characteristic and Real Intensity of Exercise in a Hospital-based Physical Activity Protocol for Patients With Chronic Disease
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Edem ALLADO, ACC-AHU, Central Hospital, Nancy, France
Other Study IDs: 2021-PI191
Record Dates: First submitted 2021-11-09; First posted 2021-12-06 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Physical Inactivity
Keywords: Adapted Physical activity; Chronic disease; exercise
MeSH Terms: conditions — Sedentary Behavior; Chronic Disease; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No limitation of exercise performance capacities: normal maximal oxygen uptake (greater than or equal to 80% of the reference value)
  Interventions: Other: Heart Rate Recording
- Limitation of exercise performance capacities: reduced maximal oxygen uptake (less than 80% of the reference value).
  Interventions: Other: Heart Rate Recording

INTERVENTIONS:
Other: Heart Rate Recording — During the APA session, HR was digitized at 1Hz (using custo guard, Custo Med GmbH). The ratio between the APA session HR and exercise test HRpeak was used to assess the intensity of effort.

SUMMARY:
The objective is to better characterize an adapted physical activity (APA) program within of the management of chronic diseases.

In France, since 2016, medical doctors have been able to prescribe APA to their patients with chronic diseases but while there are indeed prescription recommendations, there is no clear characterization of the practical reality of APA programs.

The interest of this work is to benefit from the experience of the Center of Sports Medicine and Adapted Physical Activities in Nancy (France) specifically dedicated to the prescription and the initiation of an APA program for of patients with a chronic disease.

Thus, this work aims to determine the real intensity of the APA, the effectiveness of the assessment necessary for the dispensation of the APA and other parameters likely to modify the result of the treatment.

ELIGIBILITY:
Inclusion Criteria:

- age greater than 18 years old, with the ability to perform a cardiopulmonary exercise test

Exclusion Criteria:

* beta-blocker treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional monocentric study performed at the Nancy University Center of Sports Medicine and APA, France, between February 2020 and July 2021, in patients requiring implementation of APA.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
evaluate the real intensity level of adapted physical activity (APA). | Heart rate mean during 1 hour in the first APA Session (cross-sectional monocentric study)
  evaluate the real intensity level of exercise in a sample of patients with chronic disease involved in a hospital-based program of adapted physical activity (APA).

SECONDARY OUTCOMES:
Evaluate Six-Minute Walk Test (6-MWT) efficacity to determine physical activity capacities | 6 minutes in the first APA Session (cross-sectional monocentric study)
  evaluate Six-Minute Walk Test (6-MWT) efficacity to determine physical activity capacities for patients with chronic disease.
Evaluate sit-to-stand test (1 minute)) efficacity to determine physical activity capacities | 1 minute in the first APA Session (cross-sectional monocentric study)
  Evaluate sit-to-stand test (1 minute)) efficacity to determine physical activity capacitiesfor patients with chronic disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy., Vandœuvre-lès-Nancy, France